CLINICAL TRIAL: NCT05533177
Title: Effect Analysis of Physical Therapy Based on Electronic Medical Record
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Qingdao Mental Health Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20220321
Record Dates: First submitted 2022-03-26; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-03

CONDITIONS: Physical Therapy
Keywords: rTMS; big data analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schizophrenia, schizotypal and delusional disorders: Patients in Shanghai Mental Health Center and Qingdao Mental Health Center; meet ICD-10 diagnosis of F20-F29 Schizophrenia、schizotypal and delusional disorders criteria and its subtype (mental examination was conducted by three levels of doctors including at least one attending physician and one chief physician in psychiatric); available relevant HIS system biochemical data; have been treated with physical therapy; age and gender is not limited.
- Mood disorders: Patients in Shanghai Mental Health Center and Qingdao Mental Health Center; meet ICD-10 diagnosis of F30-F39 Mood disorders criteria and its subtype (mental examination was conducted by three levels of doctors including at least one attending physician and one chief physician in psychiatric); available relevant HIS system biochemical data; have been treated with physical therapy; age and gender is not limited.
- Neurotic, stress-related and somatoform disorders: Patients in Shanghai Mental Health Center and Qingdao Mental Health Center; meet ICD-10 diagnosis of F40-F48 Neurotic、stress-related and somatoform disorders criteria and its subtype (mental examination was conducted by three levels of doctors including at least one attending physician and one chief physician in psychiatric); available relevant HIS system biochemical data; have been treated with physical therapy; age and gender is not limited.

SUMMARY:
WHO has reported the heavy disease burden of psychiatric disorders. Due to the unsatisfactory effect of pharmacotherapy, physical therapy has attracted extensive attention as a complementary therapy. However, few large sample real-world studies are exploring its efficacy. This study intends to explore the efficacy of physical therapy in different types of mental disorders, which is meaningful for the formulation of personalized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* age is not limited
* gender is not limited
* meets the diagnostic criteria of ICD-10 F20-F48 and its sub-categories
* has relevant HIS system data that can be utilized.
* have been treated with physical therapy

Exclusion Criteria:

* patients who did not meet the appeal diagnosis
* patients who met the above three diagnoses but had severe data loss (missing value ≥ estimated data value of 30%)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects are patients in Shanghai Mental Health Center and Qingdao Mental Health Center; meet ICD-10 diagnosis criteria of ICD-10 F20-F48 and its subtype (mental examination was conducted by three levels of doctors including at least one attending physician and one chief physician in psychiatric); available relevant HIS system biochemical data; have been treated with physical therapy; age and gender is not limited
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Times of outpatients visit of patients with different types of mental disorders treated with rTMS | At December 2022
  Based on electronic medical record (text profile), we will extract prognosis related information of patients treated with rTMS, namely, their times of outpatients visit.
Thyroid hormones changes of biochemical parameters after rTMS in patients with mental disorders | At March 2023
  Based on electronic medical record (record of examination information), we will extract all the patients' records of thyroid hormones. Then analyze the changes of these parameters after rTMS to see if these changes are related to the prognosis of patients with mental disorders.
Liver function related indexes changes of biochemical parameters after rTMS in patients with mental | At March 2023
  Base on electronic medical record (record of examination information), we will extract all the patients' records of liver function tests. Then analyze the changes of these parameters after rTMS to see if these changes are related to the prognosis of patients with mental disorders.
Duration of the whole outpatients visit of patients with different types of mental disorders treated with rTMS | At December 2022
  Based on electronic medical record (text profile), we will extract prognosis related information of patients treated with rTMS, namely, the duration of the whole outpatients visit.
Changes of status description of patients with different types of mental disorders treated with rTMS | At December 2022
  Based on electronic medical record (text profile), we will extract prognosis related information of patients treated with rTMS, namely, the changes of status description of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No